CLINICAL TRIAL: NCT05608083
Title: Healthy Relationships on the Autism Spectrum: Feasibility and Target Engagement
Brief Title: HEARTS R34 Feasibility Study, Autistic Participants
Acronym: HEARTS-R34
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Emily Rothman, Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 6800E
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Autism Spectrum Disorder
Keywords: Friendships; Dating relationships; Zoom sessions; Satisfaction
MeSH Terms: conditions — Autism Spectrum Disorder; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HEARTS NOW (Experimental): Participants in the HEARTS NOW group participants will participate in a weekly six-session online HEARTS class via Zoom about relationships.
  Interventions: Behavioral: HEARTS classes
- HEARTS LATER (Active Comparator): Participants in the HEARTS LATER group will participate in a six-week online support group via Zoom about relationships. Participants in this arm will have the option of taking the HEARTS class after the study has ended.
  Interventions: Behavioral: Online discussion group

INTERVENTIONS:
Behavioral: HEARTS classes — HEARTS teaches autistic adults about friendship and healthy dating relationships. HEARTS is 6-sessions long and meets weekly over zoom. Each session is 90 minutes long.
  Arms: HEARTS NOW
Behavioral: Online discussion group — A 90-minute discussion group will meet online weekly for 6 weeks to discuss friendships and healthy dating relationships for autistic adults.
  Arms: HEARTS LATER

SUMMARY:
The goal of this randomized clinical trial is to test whether the 6 sessions HEARTS Healthy Relationships classes increases the satisfaction that autistic adults feel about their friendships and dating relationships compared to a 6 weeks online discussion group. The 6 HEARTS sessions cover: healthy and unhealthy relationships, launching new relationships, neurohealth, meeting and reconnecting, boundaries, and healthy endings.

Participants who take part in this research study will be in this research study for three months. During this time, participants will be asked to complete two 30-minute and six 10-minute online surveys, and participate in two 20-minute interviews over Zoom.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with autism by a healthcare provider or other professional
* Willing to be randomized to either HEARTS or the active control condition (ACC)
* Have not already participated in the study, nor in the HEARTS class previously
* English speaking

Exclusion Criteria:

* unwilling or unable to provide informed consent by themselves
* have participated at any time previously in HEARTS research or the HEARTS class
* are unable to understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change in engaging in perspective-taking related to rejection at 6 weeks | baseline, 6 weeks
  The 25-item Host Access Table (HAT) scale self-report measure that assesses participants' ability to engage in perspective-taking related to perceived rejection and the extent to which they attribute hostile intentions to a person given an ambiguous situation will be used to measure this outcome. completed by participant. For each item participants will select either: often, sometimes, or never. Higher scores are associated with higher levels of perceived rejection.
Change in engaging in perspective-taking related to rejection at 12 weeks | baseline, 12 weeks
  The 25-item Host Access Table (HAT) scale self-report measure that assesses participants' ability to engage in perspective-taking related to perceived rejection and the extent to which they attribute hostile intentions to a person given an ambiguous situation will be used to measure this outcome. completed by participant. For each item participants will select either: often, sometimes, or never. Higher scores are associated with higher levels of perceived rejection.
Change in resilience capacity given social rejection at 6 weeks | baseline, 6 weeks
  The Rejection Sensitivity Questionnaire (RSQ), a 10-item self-report measure that assesses participants' capacity to be resilient when experiencing social rejection such as sending a text message and not getting a reply, will be used to assess this outcome. Lower scores are associated with more resilience given rejection.
Change in resilience capacity given social rejection at 12 weeks | baseline, 12 weeks
  The Rejection Sensitivity Questionnaire (RSQ), a 10-item self-report measure that assesses participants' capacity to be resilient when experiencing social rejection such as sending a text message and not getting a reply, will be used to assess this outcome. Lower scores are associated with more resilience given rejection.
Change in satisfaction with close relationships at 6 weeks | baseline, 6 weeks
  The Clinical Global Impressions-Severity/Improvement (CGI-S/I), a global measure of improvement and functioning, will be used to measure satisfaction with quality of close relationships. Each of the 3 items are rated on a 7-point scale from: 1 (normal) to 7 (amongst the most severely ill patients). CGI-C scores range from 1 (very much improved) through to 7 (very much worse). Lower scores are favorable.
Change in satisfaction with close relationships at 12 weeks | baseline, 12 weeks
  The Clinical Global Impressions-Severity/Improvement (CGI-S/I), a global measure of improvement and functioning, will be used to measure satisfaction with quality of close relationships. Each of the 3 items are rated on a 7-point scale from: 1 (normal) to 7 (amongst the most severely ill patients). CGI-C scores range from 1 (very much improved) through to 7 (very much worse). Lower scores are favorable.
Change in motivation to interact socially at 6 weeks | baseline, 6 weeks
  The semi-structured social motivation interview (SMI) will be conducted by an independent evaluator to assess internal cognition related to desire, interest, and behaviors reflective of degree of motivation to interact socially.
Change in motivation to interact socially at 12 weeks | baseline, 12 weeks
  The semi-structured social motivation interview (SMI) will be conducted by an independent evaluator to assess internal cognition related to desire, interest, and behaviors reflective of degree of motivation to interact socially.

SECONDARY OUTCOMES:
Participant satisfaction with study participation | 12 weeks
  An investigator developed 2-item assessment will be used to assess participants' feelings about the research-related consent procedure, and experiences with the research team. Participants will indicate their satisfaction on a scale from 1 to 10, where 10 represents highest satisfaction.
Participant feelings of acceptability of study intervention | 12 weeks
  An investigator developed self report 3-item scale to assess participants' feelings about whether HEARTS was informative, interesting, how likely participants would be to recommend it to other people and suggestions for how it could be improved will be used to assess this outcome. Participants will indicate their satisfaction on a scale from 1 to 10, where 10 represents highest satisfaction.
Participant rating of content acceptability | weekly during the 6 weeks of the interventions
  This outcome will be assessed by self reported ratings on each piece of intervention content after each class session, indicating how useful participants found the content. Participants will indicate their satisfaction with usefulness on a scale from 1 to 10, where 10 represents highest satisfaction.
Teacher rating of participant engagement and satisfaction | weekly during the 6 weeks of the interventions
  Teachers of the HEARTS intervention will complete a 3-item survey to assess their rating of participant engagement and satisfaction scores (PESS). Scores can range from 0 to 3 where 0 is low and 3 is high satisfaction. Higher scores are more favorable.

CONTACTS AND LOCATIONS:
Overall Officials: Emily F Rothman, ScD, Principal Investigator — BU Sargent College, Occupational Therapy Department
Locations (1):
- Boston University CRC, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No